CLINICAL TRIAL: NCT04157179
Title: Cerebral Oxygen Metabolism in Children
Acronym: COMIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 201905044
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Sickle Cell Disease; Cerebral Stroke
Keywords: extracorporeal membrane oxygenation; cerebrovascular reactivity; sickle cell disease; healthy controls; magnetic resonance imaging
MeSH Terms: conditions — Anemia, Sickle Cell; Stroke | interventions — Carbon Dioxide

STUDY DESIGN:
Intervention Model Description: All arms will receive the same study conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy Controls (Active Comparator)
  Interventions: Other: Carbon Dioxide
- Extracorporeal Membrane Oxygenation survivors (Active Comparator)
  Interventions: Other: Carbon Dioxide
- Sickle Cell Anemia participants (Active Comparator)
  Interventions: Other: Carbon Dioxide

INTERVENTIONS:
Other: Carbon Dioxide — Participants inhale carbon dioxide while in magnetic resonance imaging scan to measure cerebrovascular reactivity

SUMMARY:
The purpose of this research study is to better understand how blood flow and metabolism change can influence brain development in the early decades of life.

We will examine brain blood flow and metabolism using magnetic resonance imaging (MRI). The brain's blood vessels expand and constrict to regulate blood flow based on the brain's needs. The amount of expanding and contracting the blood vessels can do varies by age. The brain's blood flow changes in small ways during everyday activities, such as normal brain growth, exercise, or deep concentration. Significant illness or psychological stress may increase the brain's metabolic demand or cause other bigger changes in blood flow. If blood vessels are not able to expand to give more blood flow when metabolic demand is high, the brain may not get all of the oxygen it needs. In extreme circumstances, if the brain is unable to get enough oxygen for a long time, a stroke may occur. Sometimes small strokes occur without other noticeable changes and are only detectable on an MRI. These are sometimes called "silent strokes." In less extreme circumstances, not having as much oxygen as it wants may cause the brain to grow and develop more slowly than it should.

One way to test the ability of blood vessels to expand is by measuring blood flow while breathing in carbon dioxide. Carbon dioxide causes blood vessels in the brain to dilate without increasing brain metabolism.

During this study participants may be asked to undergo a blood draw, MRI, and potential neuropsychological assessments. It is also possible that the study team will use a special mask to control the amount of carbon dioxide the participants breathe in so they don't breathe in too much.

DETAILED DESCRIPTION:
The purpose of the study is to identify imaging biomarkers for brain tissue under high metabolic stress at risk for permanent injury. We will measure CBF, OEF, and CVR in children with and without perturbations in cerebral oxygen delivery over time to determine each parameter's role in clinical and radiologic neurologic outcomes. Measuring CBF and OEF can be done with specialized MRI sequences. Measuring CVR requires a vasoactive response, such as carbon dioxide. In order to delivery carbon dioxide evenly and as safely as possible, we will use an MRI-compatible device to prevent over-breathing carbon dioxide and allow rapid steady-state physiology to minimize total scan time.

ELIGIBILITY:
Healthy Controls:

* Healthy controls ages 3-50 years of age
* Able to participate in MRI scan without sedation
* Not currently pregnant
* No significant psychiatric history, defined as having a severe psychiatric diagnosis, per PI discretion
* No history of epilepsy
* No history of stroke or cerebrovascular disease
* May have occasional headaches if not taking a daily preventative medication for headaches
* Not on vasodilatory medication, such as sildenafil or verapamil

Sickle Cell Anemia Participants:

* Ages 3-50 years of age
* Hb SS or SBeta-thal
* Able to participate in MRI scan without sedation
* Not currently pregnant
* Not on vasodilatory medication, such as sildenafil or verapamil

Extracorporeal Membrane Oxygenation (ECMO) Survivors:

* Ages 3-50 years of age
* History of cannulation for ECMO
* Able to participate in MRI scan without sedation
* Not currently pregnant
* Not on vasodilatory medication, such as sildenafil or verapamil

Ages: 3 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 350 (Estimated)
Dates: Start 2019-10-17 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Cerebral Oxygen Metabolism | From the beginning of the MRI scan to the completion of the MRI scan -- 75 minutes.

SECONDARY OUTCOMES:
Cerebrovascular Reactivity | From administration of carbon dioxide to end of inhalation of carbon dioxide -- 15 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University of St. Louis, St Louis, Missouri, United States